CLINICAL TRIAL: NCT00001595
Title: A Clinical and Genetic Investigation of Pituitary and Hypothalamic Tumors and Related Disorders
Brief Title: An Investigation of Pituitary Tumors and Related Hypothalmic Disorders
Status: Recruiting | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 970076; 97-CH-0076
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-01-16

CONDITIONS: Panhypopituitarism; Gigantism/Acromegaly; Prolactinoma; Cushing Disease
Keywords: Developmental Defect; Oncogenesis; Evaluation and Management; Psychological; Cushing Disease; Natural History
MeSH Terms: conditions — Combined Pituitary Hormone Deficiency; Gigantism; Acromegaly; Prolactinoma; Pituitary ACTH Hypersecretion; Congenital Abnormalities; Carcinogenesis | interventions — Tissue Banks

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with pituitary tumors or hypothalmic defects: Patients with pituitary tumors or hypothalmic defects
  Interventions: Procedure: MRI; Procedure: Tissue specimen collection

INTERVENTIONS:
Procedure: MRI
Procedure: Tissue specimen collection

SUMMARY:
There is a variety of tumors affecting the pituitary gland in childhood; some of these tumors (eg craniopharyngioma) are included among the most common central nervous system tumors in childhood. The gene(s) involved in the pathogenesis of these tumors are largely not known; their possible association with other developmental defects or inheritance pattern(s) has not been investigated. The present study serves as a (i) screening/training, and, (ii) a research protocol.

As a screening and training study, this protocol allows our Institute to admit children with tumors of the hypothalamic-pituitary unit to the pediatric endocrine clinics and wards of the NIH Clinical Center for the purposes of

(i) training our fellows and students in the identification of genetic defects associated with pituitary tumor formation, and

(ii) teaching our fellows and students the recognition, management and complications of pituitary tumors

As a research study, this protocol aims at

(i) developing new clinical studies for the recognition and therapy of pituitary tumors; as an example, two new studies have emerged within the context of this protocol: (a) investigation of a new research magnetic resonance imaging (MRI) tool and its usefulness in the identification of pituitary tumors, and (b) investigation of the psychological effects of cortisol secretion in pediatric patients with Cushing disease. Continuation of this protocol will eventually lead to new, separate protocols that will address all aspects of diagnosis of pituitary tumors and their therapy in childhood.

(ii) Identifying the genetic components of pituitary oncogenesis; those will be investigated by (a) studying the inheritance pattern of pituitary tumors in childhood and their possible association with other conditions in the families of the patients, and (ii) collecting tumor tissues and examining their molecular genetics. As with the clinical studies, the present protocol may help generate ideas for future studies on the treatment and clinical follow up of pediatric patients with tumors of the pituitary gland and, thus, lead to the development of better therapeutic regimens for these neoplasms....

DETAILED DESCRIPTION:
Study Description:<TAB>

This protocol aims to evaluate subjects with tumors of the hypothalamic pituitary unit to: identify genetic components of pituitary and hypothalamic oncogenesis, to develop new clinical studies for the recognition and therapy of pituitary tumors, and to investigate the psychological effects of cortisol secretion.

Objectives:<TAB>

Primary Objective:

To collect peripheral blood samples and tumor tissues and examine the molecular genetics of the specimens, in an effort to elucidate developmental pathways leading to pituitary gland oncogenesis and/or other defects.

Secondary Objectives:

To serve as a screening protocol for future studies on the treatment and clinical follow up of our patients with pituitary tumors; it is our hope that the protocol will continue to be a vehicle for the development of more related clinical studies.

To collect biospecimens.

To evaluate the cognitive, psychological, and patient-reported health status of mental and social well-being and symptoms of hypercortisolemia and adrenal insufficiency (AI) associated with recovery from Cushing syndrome (CS) in children with this disease.

Endpoints:

<TAB>

Primary Endpoint:

Molecular genetic testing

Secondary Endpoints:

Pre- and/or post- treatment assessment of research variables related to pituitary/hypothalamic tumors and comorbidities.

Cognitive, behavioral, psychological, and patient-reported outcomes

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Stated willingness to comply with all study procedures and availability for the duration of the study.
2. Male or female with:

   1. Evidence for the existence of a tumor of the hypothalamic-pituitary unit or related disorder, as indicated by previously obtained imaging studies or biochemical investigation of the hypothalamo-hypophyseal function (aged 2 years to 70 years)

      or
   2. Family members (any age) of patients with a family history of tumors of the hypothalamic-pituitary unit or related disorders as part of the linkage part of the study, or
   3. Members (any age) of a kindred suspected of having an inherited form of neoplasia of the hypothalamic-pituitary unit or related disorder, as evidenced by results of a patient enrolled in this protocol, as part of the linkage part of the study
3. Ability of the subject or LAR to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Pregnancy: Pregnancy will be evaluated only in participants of reproductive age (from 10 years old until 60 years of age unless menopause has already occurred per clinical report of the participant).

   For participants enrolled as external participants or under the Linkage study (where research activities include no more than blood draws), any female who could possibly become pregnant will be screened using clinical criteria (history, with pregnancy testing only if indicated) for exclusion and this information will be documented in the consent process note in EMR. If a participant has initially been registered as external location and then presents on-site, then pregnancy test will be performed if within the reproductive age group.
2. Patients with any medical, physical, psychiatric, or social condition, which, in the opinion of the investigators, would make participation in this protocol not in their best interest, will be excluded from the study.
3. Patients who are critically ill, unstable, or with severe organ failure that may affect/limit the endocrine evaluation and place unsustainable demands on CC or NICHD resources may be excluded.

Ages: 2 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects with known or suspected pituitary or hypothalamic tumors or related disorders. Family members (adult and pediatric; affected and unaffected) may be enrolled in the DNA linkage analysis part of this protocol.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 1997-04-21 (Actual)

PRIMARY OUTCOMES:
Molecular genetic testing, whole exome sequencing | ongoing
  To collect peripheral blood samples and tumor tissues and examine the molecular genetics of the specimens, in an effort to elucidate developmental pathways leading to pituitary gland oncogenesis and/or other defects.

SECONDARY OUTCOMES:
To investigate the usefulness of a new MRI of the pituitary gland | completed
  Comparison of MRI techniques to identify micro adenomas
To identify the clinical and genetic features of pituitary tumors by investigating their inheritance pattern and possible association with other conditions in the families of the patients. | ongoing
  Genetic studies of pituitary and hypothalamic tumors or related disorders
To evaluate the cognitive, psychological, and patient-reported health status of mental and social well-being and symptoms of adrenal insufficiency associated with Cushing syndrome in children with this disease. | ongoing
  Descriptive study of cognitive, psychological, and patient-reported health status of mental and social well-being associated with Cushing and after treatment
To collect peripheral blood samples and tumor tissues and examine the molecular genetics of the specimens, in an effort to elucidate developmental pathways leading to pituitary gland oncogenesis and/or other defects | ongoing
  Genetic studies of pituitary and hypothalamic tumors or related disorders

CONTACTS AND LOCATIONS:
Overall Officials: Deborah P Merke, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified Samples/data, including genomic data, will be shared with NIH & non-NIH collaborators after an MTA is obtained. If coded data shared, the key code will not be shared with collaborators & stay at NIH. If Data & samples shared with AIs and IC with an FWA/operating under the DOH and reported at the time of CR. Sharing with AIs without an FWA/operating under the DoH will be submitted for prospective IRB approval. Submissions to NIH-sponsored or supported databases and repositories will be reported at the time of CR. Submission to non-NIH sponsored or supported databases & repositories will be submitted for prospective IRB approval.@@@@@@Required approvals from the collaborating institution will be obtained and materials will be shipped in accordance with NIH and federal regulations. This study will comply with the NIH GDS Policy, which applies to all NIH-funded research that generates large-scale human or non-human GD, as well as the use of these data for subsequent research.
Supporting Information: Study Protocol
Time Frame: AIs in the NIH intramural program may participate with NIH/ non-NIH collaborators under which de-identified human materials are transferred from the intramural program to another site for correlative studies that are part of the approved protocol. In this case, the protocol clearly documents the tests conducted under the correlative studies& each institution participating in the clinical study is bound by the terms of this Protocol& their obligations under the statutes & regulations. @@@@@@This study will comply with the NIH DSP &Policy on the Dissemination of NIH-Funded CT Information & Registration & Results Information Submission rule. As such, this trial will be registered at CT.gov,& results information from this trial will be submitted to CT.gov. In addition, every attempt will be made to publish results in peer-reviewed journals. Data from this study may be requested from other researchers 3 years after the completion of the primary endpoint by contacting PI or NICHD-DASH.
Access Criteria: This study will comply with the NIH Data Sharing Policy and Policy on the Dissemination of NIH-Funded Clinical Trial Information and the Clinical Trials Registration and Results Information Submission rule. As such, this trial will be registered at ClinicalTrials.gov, and results information from this trial will be submitted to ClinicalTrials.gov. In addition, every attempt will be made to publish results in peer-reviewed journals. Data from this study may be requested from other researchers 3 years after the completion of the primary endpoint by contacting PI or NICHD-DASH.

REFERENCES:
- [Background] Trivellin G, Daly AF, Faucz FR, Yuan B, Rostomyan L, Larco DO, Schernthaner-Reiter MH, Szarek E, Leal LF, Caberg JH, Castermans E, Villa C, Dimopoulos A, Chittiboina P, Xekouki P, Shah N, Metzger D, Lysy PA, Ferrante E, Strebkova N, Mazerkina N, Zatelli MC, Lodish M, Horvath A, de Alexandre RB, Manning AD, Levy I, Keil MF, Sierra Mde L, Palmeira L, Coppieters W, Georges M, Naves LA, Jamar M, Bours V, Wu TJ, Choong CS, Bertherat J, Chanson P, Kamenicky P, Farrell WE, Barlier A, Quezado M, Bjelobaba I, Stojilkovic SS, Wess J, Costanzi S, Liu P, Lupski JR, Beckers A, Stratakis CA. Gigantism and acromegaly due to Xq26 microduplications and GPR101 mutation. N Engl J Med. 2014 Dec 18;371(25):2363-74. doi: 10.1056/NEJMoa1408028. Epub 2014 Dec 3. PMID 25470569
- [Background] Stratakis CA, Carney JA, Lin JP, Papanicolaou DA, Karl M, Kastner DL, Pras E, Chrousos GP. Carney complex, a familial multiple neoplasia and lentiginosis syndrome. Analysis of 11 kindreds and linkage to the short arm of chromosome 2. J Clin Invest. 1996 Feb 1;97(3):699-705. doi: 10.1172/JCI118467. PMID 8609225
- [Background] Magiakou MA, Mastorakos G, Oldfield EH, Gomez MT, Doppman JL, Cutler GB Jr, Nieman LK, Chrousos GP. Cushing's syndrome in children and adolescents. Presentation, diagnosis, and therapy. N Engl J Med. 1994 Sep 8;331(10):629-36. doi: 10.1056/NEJM199409083311002. PMID 8052272
- [Derived] Trivellin G, Sanchez-Gaya V, Grasso A, Pasinska M, Stratakis CA, Milnes D, Kirk EP, Beckers A, Lania AG, Petrossians P, Rada-Iglesias A, Franke M, Daly AF. Distinguishing benign from pathogenic duplications involving GPR101 and VGLL1-adjacent enhancers in the clinical setting with the bioinformatic tool POSTRE. NPJ Genom Med. 2026 Jan 15. doi: 10.1038/s41525-025-00548-7. Online ahead of print. PMID 41540017
- [Derived] Omotosho YB, Reynolds JC, Yanovski JA, Tatsi C. Body Composition and Fat Deposition in Children with Cushing Disease and Associations with Cardiometabolic Risk Factors. J Pediatr. 2025 Dec 3;290:114933. doi: 10.1016/j.jpeds.2025.114933. Online ahead of print. PMID 41349930
- [Derived] Zainab R, Kaur S, Lack J, Similuk M, Tandon M, Ghosh R, Seifert BA, Tokita M, Flippo C, Yan J, Walkiewicz M, Chittiboina P, Tatsi C. Genetic evaluation of pediatric pituitary adenomas and USP8-related genotype-phenotype correlations in Cushing's disease. Pituitary. 2025 Aug 14;28(5):92. doi: 10.1007/s11102-025-01557-6. PMID 40813536
- [Derived] Hernandez-Ramirez LC, Pankratz N, Lane J, Faucz FR, Chittiboina P, Kay DM, Beethem Z, Mills JL, Stratakis CA. Genetic drivers of Cushing's disease: Frequency and associated phenotypes. Genet Med. 2022 Dec;24(12):2516-2525. doi: 10.1016/j.gim.2022.08.021. Epub 2022 Sep 23. PMID 36149413
- [Derived] Martinez de LaPiscina I, Hernandez-Ramirez LC, Portillo N, Gomez-Gila AL, Urrutia I, Martinez-Salazar R, Garcia-Castano A, Aguayo A, Rica I, Gaztambide S, Faucz FR, Keil MF, Lodish MB, Quezado M, Pankratz N, Chittiboina P, Lane J, Kay DM, Mills JL, Castano L, Stratakis CA. Rare Germline DICER1 Variants in Pediatric Patients With Cushing's Disease: What Is Their Role? Front Endocrinol (Lausanne). 2020 Jul 3;11:433. doi: 10.3389/fendo.2020.00433. eCollection 2020. PMID 32714280
- [Derived] Chasseloup F, Pankratz N, Lane J, Faucz FR, Keil MF, Chittiboina P, Kay DM, Hussein Tayeb T, Stratakis CA, Mills JL, Hernandez-Ramirez LC. Germline CDKN1B Loss-of-Function Variants Cause Pediatric Cushing's Disease With or Without an MEN4 Phenotype. J Clin Endocrinol Metab. 2020 Jun 1;105(6):1983-2005. doi: 10.1210/clinem/dgaa160. PMID 32232325
- [Derived] Hodes A, Meyer J, Lodish MB, Stratakis CA, Zilbermint M. Mini-review of hair cortisol concentration for evaluation of Cushing syndrome. Expert Rev Endocrinol Metab. 2018 Sep;13(5):225-231. doi: 10.1080/17446651.2018.1517043. Epub 2018 Sep 20. PMID 30234410
- [Derived] Saldarriaga C, Lyssikatos C, Belyavskaya E, Keil M, Chittiboina P, Sinaii N, Stratakis CA, Lodish M. Postoperative Diabetes Insipidus and Hyponatremia in Children after Transsphenoidal Surgery for Adrenocorticotropin Hormone and Growth Hormone Secreting Adenomas. J Pediatr. 2018 Apr;195:169-174.e1. doi: 10.1016/j.jpeds.2017.11.042. Epub 2018 Feb 1. PMID 29395172
- [Derived] Birdwell L, Lodish M, Tirosh A, Chittiboina P, Keil M, Lyssikatos C, Belyavskaya E, Feelders RA, Stratakis CA. Coagulation Profile Dynamics in Pediatric Patients with Cushing Syndrome: A Prospective, Observational Comparative Study. J Pediatr. 2016 Oct;177:227-231. doi: 10.1016/j.jpeds.2016.06.087. Epub 2016 Aug 2. PMID 27496264
- [Derived] Gourgari E, Lodish M, Keil M, Wesley R, Hill S, Xekouki P, Lyssikatos C, Belyavskaya E, De La Luz SM, Stratakis CA. Post-operative growth is different in various forms of pediatric Cushing's syndrome. Endocr Relat Cancer. 2014;21(6):L27-31. doi: 10.1530/ERC-14-0405. Epub 2014 Sep 25. No abstract available. PMID 25258026
- [Derived] Lodish MB, Gourgari E, Sinaii N, Hill S, Libuit L, Mastroyannis S, Keil M, Batista DL, Stratakis CA. Skeletal maturation in children with Cushing syndrome is not consistently delayed: the role of corticotropin, obesity, and steroid hormones, and the effect of surgical cure. J Pediatr. 2014 Apr;164(4):801-6. doi: 10.1016/j.jpeds.2013.11.065. Epub 2014 Jan 10. PMID 24412141
- [Derived] Keil MF, Graf J, Gokarn N, Stratakis CA. Anthropometric measures and fasting insulin levels in children before and after cure of Cushing syndrome. Clin Nutr. 2012 Jun;31(3):359-63. doi: 10.1016/j.clnu.2011.11.007. Epub 2011 Dec 7. PMID 22154461
- [Derived] Keil MF, Stratakis CA. Facial metrics in children with corticotrophin-producing pituitary adenomas suggest abnormalities in midface development. J Pediatr Endocrinol Metab. 2009 Jan;22(1):47-53. doi: 10.1515/jpem.2009.22.1.47. PMID 19344074
- [Derived] Keil MF, Merke DP, Gandhi R, Wiggs EA, Obunse K, Stratakis CA. Quality of life in children and adolescents 1-year after cure of Cushing syndrome: a prospective study. Clin Endocrinol (Oxf). 2009 Sep;71(3):326-33. doi: 10.1111/j.1365-2265.2008.03515.x. Epub 2008 Dec 17. PMID 19170709
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1997-CH-0076.html